CLINICAL TRIAL: NCT00919932
Title: Using a Text-message System to Engage Depressed Adolescents in Cognitive-behavioral Therapy Homework.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Han-chun Liang, Resident Physician, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACA-08-001-UPMC
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Major Depressive Disorder; Cognitive Behavior Therapy; Text Messaging
Keywords: Depression; CBT; Texting; SMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paper and pen homework (Active Comparator): Treatment as usual: therapy homework is completed by paper and pen.
  Interventions: Behavioral: Paper and pen homework
- Text-message homework (Experimental): Experimental treatment: therapy homework is completed by text messaging.
  Interventions: Device: Text message system homework.

INTERVENTIONS:
Behavioral: Paper and pen homework — Homework will be standardized through the use of Judith Beck's dysfunctional thought record (DTR), which is a primary tool for patients to evaluate and respond in writing to their automatic thoughts (Beck 126). The homework will be done on a preprinted form which is assigned weekly and reviewed with their therapists at weekly sessions for 4 weeks.
  Arms: Paper and pen homework
Device: Text message system homework. — Homework will be standardized through the use of Judith Beck's dysfunctional thought record (DTR), which is a primary tool for patients to evaluate and respond in writing to their automatic thoughts (Beck 126). The novel text-messaging system allows homework to be submitted directly through an adolescent's cellular phone, includes text-messaged homework reminder prompts, and collates all homework for therapists to review with patients during therapy sessions. This is assigned and reviewed weekly for 4 weeks.
  Arms: Text-message homework

SUMMARY:
The primary goal of the pilot is to test the feasibility and utility of using a text-messaging system to engage adolescents in improved homework adherence during cognitive-behavioral therapy (CBT) for major depressive disorder.

DETAILED DESCRIPTION:
Adolescent major depressive disorder leads to recurrent episodes, increased rates of attempted and completed suicides, and persistent social impairment between episodes (Weissman et al 1999). Cognitive behavioral therapy (CBT) is an accepted first-line therapy for mild-moderate depression in adolescents. Integral to CBT is "homework" as it enhances mastery of newly learned coping strategies, facilitates generalization of skills to novel situations, increases self-efficacy, and ultimately reduces vulnerability to relapse (Detweiler et al 1999). Adherence to homework is a recognized problem in adults, and is similarly problematic in adolescents. One method of implementing CBT homework in a manner that is centric to current youth culture is through text messaging. By using a modern modality that many adolescents rely on for daily communication, there is the likelihood that they will find it more engaging than traditional modalities. Thus the potential that a text message system can help improve homework compliance in adolescents is significant, because improved homework adherence may ultimately be linked to improved clinical outcomes for these disorders with high rates of chronic morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder
* own a cellular phone with text messaging capabilities

Exclusion Criteria:

* history of psychosis
* history of mental retardation
* active suicidal ideation or intent

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han-chun Liang, MD, Principal Investigator — University of Pittsburgh

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paper and Pen Homework | Text-message Homework
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paper and Pen Homework | Text-message Homework | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Therapy Homework Compliance: Percent Homework Completed
Description: Number of thought logs completed over the course of the 4 week trial.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: homework sheets completed
Arm/Group | Paper and Pen Homework | Text-message Homework
Number analyzed (Participants) | 4 | 5
homework sheets completed
  Week 1 | .44 (0.27) | 0 (0)
  Week 2 | 0.47 (0.39) | 0.25 (0.4)
  Week 3 | 0.37 (0.35) | 0 (0)
  Week 4 | 0.27 (0.24) | 0 (0)

2. Secondary Outcome: Exit Interview
Description: Verbal interview
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Paper and Pen Homework | Text-message Homework
Number analyzed (Participants) | 4 | 5
participants | 4 | 5

ADVERSE EVENTS:
Arm/Group | Paper and Pen Homework | Text-message Homework
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No